CLINICAL TRIAL: NCT04883164
Title: Immunity After COVID-19 Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Plexision (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00053511
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Immunity to COVID-19
MeSH Terms: interventions — Cell Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples, White blood cells extracted from whole blood samples, serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy non-immunocompromized subjects: Healthy individuals are those with no pre-existing conditions that cause immune deficiency, and who are not receiving drugs to suppress the immune system.
  •
  Interventions: Other: Cellular and antibody response to spike antigens of SARS-CoV-2 in both groups in peripheral blood samples
- Immunocompromized: Immunocompromised subjects are those receiving immunosuppressive or immunomodulatory drugs such as those given for autoimmune disease, inflammatory bowel disease, malignancies and transplantation. Bone marrow transplant recipients and subjects with known immune deficiency diseases are also considered immunocompromised.
  Interventions: Other: Cellular and antibody response to spike antigens of SARS-CoV-2 in both groups in peripheral blood samples

INTERVENTIONS:
Other: Cellular and antibody response to spike antigens of SARS-CoV-2 in both groups in peripheral blood samples — Cellular immunity will be assessed with T-cells and other immune cells that express CD154 or other inflammatory or other markers after stimulation with spike antigens. Antibody immunity will be measured with binding and neutralizing activity of antibodies to spike antigens.

SUMMARY:
The purpose of the research is to evaluate new blood tests, which measure immunity to the COVID-19 coronavirus after vaccination. These tests will be used to measure T-cell and antibody immunity after COVID-19 vaccination. Recent studies show that less than one-fifth of chronically immunosuppressed transplant recipients developed anti-receptor-binding domain antibodies after the first dose of the Pfizer vaccine (Boyarski, 2021).

ood sampling at periodic intervals. These samples will be used to measure T-cell and antibody immunity to the COVID-19 coronavirus.

DETAILED DESCRIPTION:
Study type: Open-label, prospective, non-randomized, observational study.

Risk level. Minimal risk.

Blood sampling: 10 ml each time, up to 8 times in 12 month study period for each subject, minimum interval between samples is 2 weeks.

Measurements: T-cells responsive to the spike antigens of SARS-CoV-2 will be measured with flow cytometry. Antibodies specific for spike antigenic sequences will be measured with ELISA.

Inclusion criteria:

* IRB-approved informed consent,
* age 18 years or older, male or female,
* anyone considering COVID-19 vaccination or anyone that has received COVID-19 vaccination.
* Subjects can enroll at anytime after vaccination even though they may not have enrolled before vaccination.
* For individuals previously tested at Plexision for other purposes, and who have since been vaccinated, residual cells stored for quality control and potential repeat testing will be used to establish earlier measurement of cellular and antibody immunity .

Exclusion: Failure to provide informed consent

Sampling Frequency and timing: Up to 8 total samples in 12 months, 10 ml per sample, no sample to be obtained less than 2 weeks after preceding sample. Samples will be obtained

* Before vaccination
* Two to four weeks after the first dose of mRNA vaccines, or after the final dose of non-mRNA vaccines which may only require a single dose
* Two to four weeks after the second dose of the mRNA vaccines.
* Month 2 after the final dose of non-mRNA vaccine which is given only once
* 3-monthly after the first vaccine dose until month 12.

Planned enrollment: 300 total patients at least half of whom are immunocompromized.

Immunocompromized patients include but are not limited to those receiving immunosuppressive or immunomodulatory drugs such as those given for autoimmune disease, inflammatory bowel disease, malignancies and transplantation. Bone marrow transplant recipients and subjects with known immune deficiency diseases are also considered immunocompromised.

ELIGIBILITY:
Inclusion Criteria:

* IRB-approved informed consent,
* age 18 years or older, male or female,
* anyone considering COVID-19 vaccination or anyone that has received COVID-19 vaccination.
* Subjects can enroll at anytime after vaccination even though they may not have enrolled before vaccination.
* For individuals previously tested at Plexision for other purposes, and who have since been vaccinated, residual cells stored for quality control and potential repeat testing will be used to establish earlier measurement of cellular and antibody immunity as described in Table 1.

Exclusion Criteria:

* Failure to provide informed consent

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects age 18 years or older, male or female, • anyone considering COVID-19 vaccination or anyone that has received COVID-19 vaccination. • Subjects can enroll at anytime after vaccination even though they may not have enrolled before vaccination.
  * For individuals previously tested at Plexision for other purposes, and who have since been vaccinated, residual cells stored for quality control and potential repeat testing will be used to establish earlier measurement of cellular and antibody immunity.
  * Medication history such as immunosuppressive or immune modulatory drugs that are being used,
  * Underlying conditions related to immunosuppressive or immunomodulatory drug use, type of COVID-19 vaccine and doses received at the time of enrollment.
  * Other underlying conditions such as diabetes, hypertension and asthma.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
T-cells and other immune cells reactive to the spike antigenic protein and its components | 2 years
  as above, will be measured with flow cytometry
Binding and neutralizing antibodies to the spike protein and its earlier compoent | 2 years
  Antibodies will be measured by ELISA

SECONDARY OUTCOMES:
COVID-19 infection | 2 years
  diagnosed with PCR

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Reddy, BE, Principal Investigator — Plexision
Locations (1):
- Plexision, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Plexision offers antibody testing of IgG to RBD and spike proteins as clinical tests to look for infection status. Because these tests are being used to perform antibody immunity testing after vaccination in this study, Plexision will inform participants about results of this testing as they become available.